CLINICAL TRIAL: NCT05181696
Title: Radiographic Severity Scoring System and Clinical and Laboratory Evolution of COVID-19 Pneumonia
Brief Title: Retrospective Analysis of Chest X-ray Severity Scoring System of COVID-19 Pneumonia
Acronym: RANCH-COVID
Status: Recruiting | Type: Observational
Sponsor: Osijek University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OsijekUH-RC
Record Dates: First submitted 2022-01-04; First posted 2022-01-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: COVID-19 Pneumonia; Sepsis; SARS-CoV-2 Acute Respiratory Disease; Pneumonia; Multiorgan Failure
Keywords: COVID-19; Acute respiratory distress syndrome (ARDS); Sepsis; Multiorgan Failure; Chest X-ray; Inflammation
MeSH Terms: conditions — Sepsis; Pneumonia; Multiple Organ Failure; COVID-19; Respiratory Distress Syndrome; Inflammation | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 pneumonia patients: Patients treated at the University Hospital Osijek Respiratory Center with pneumonia caused by SARS-CoV-2
  Interventions: Diagnostic Test: Chest X-ray

INTERVENTIONS:
Diagnostic Test: Chest X-ray — Retrospective analysis of chest x-rays of patients with COVID-19

SUMMARY:
The research will be retrospective, and will include all patients who were admitted during 2020 and 2021 in the COVID-19 ICU of University Hospital Center Osijek due to pneumonia caused by the Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The association of chest x-ray infiltrate evolution with changes in laboratory inflammatory parameters and respiratory function parameters will be examined.

DETAILED DESCRIPTION:
The research will be retrospective, and will include a review of medical history of all patients admitted in the COVID-19 ICU of the University hospital Osijek during 2020 and 2021. Associated comorbidity, hospital admission date, intubation date, mechanical ventilation, extubation, discharge, and patient final outcome will be recorded for each patient. By analyzing X-rays of the lungs by radiology specialists, inflammatory infiltrates in the lungs will be quantified via the Brixia system, during hospital admission, admission to the Respiratory Center, and during treatment at the Respiratory Center. All patients will have their Sequential Organ Failure Assessment (SOFA) and/or Acute Physiology and Chronic Health Evaluation (APACHE II) values calculated upon admission. Inflammatory parameters (c-reactive protein (CRP), procalcitonin (PCT), interleukine-6 (IL-6), ferritin), red blood cell count, leukocytes, blood urea nitrogen (BUN), arterial blood gases and ventilation parameters on admission to the hospital, admission to the ICU, and on several occasions during treatment in the ICU will be analysed. Also, empirical use of antibiotics, the occurrence of bacterial superinfections, sepsis and organic failure will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Pneumonia caused by SARS-CoV-2 virus
* Admission to the ICU COVID-19 unit

Exclusion Criteria:

- Patients with lung tumors or history of lung resection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated in ICU COVID-19 with a diagnosis of pneumonia will be analyzed retrospectively.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Chest x-ray severity score | 21 days
  The influence of the dynamics of radiographic changes quantified by Brixia score on the outcome of COVID-19 patients will be examined
Inflammatory markers | 21 days
  The influence of serum levels of inflammatory parameters, and clinical and laboratory indicators of organic failure on chest x-ray severity score will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Nenad Nešković, PhD, Principal Investigator — University Hospital Osijek
Locations (1):
- University hospital Osijek, Osijek, Croatia

REFERENCES:
- [Background] Booth A, Reed AB, Ponzo S, Yassaee A, Aral M, Plans D, Labrique A, Mohan D. Population risk factors for severe disease and mortality in COVID-19: A global systematic review and meta-analysis. PLoS One. 2021 Mar 4;16(3):e0247461. doi: 10.1371/journal.pone.0247461. eCollection 2021. PMID 33661992
- [Background] Wolff D, Nee S, Hickey NS, Marschollek M. Risk factors for Covid-19 severity and fatality: a structured literature review. Infection. 2021 Feb;49(1):15-28. doi: 10.1007/s15010-020-01509-1. Epub 2020 Aug 28. PMID 32860214
- [Background] Mahat RK, Panda S, Rathore V, Swain S, Yadav L, Sah SP. The dynamics of inflammatory markers in coronavirus disease-2019 (COVID-19) patients: A systematic review and meta-analysis. Clin Epidemiol Glob Health. 2021 Jul-Sep;11:100727. doi: 10.1016/j.cegh.2021.100727. Epub 2021 Mar 20. PMID 33778183
- [Background] Borghesi A, Maroldi R. COVID-19 outbreak in Italy: experimental chest X-ray scoring system for quantifying and monitoring disease progression. Radiol Med. 2020 May;125(5):509-513. doi: 10.1007/s11547-020-01200-3. Epub 2020 May 1. PMID 32358689
- [Background] Borghesi A, Zigliani A, Masciullo R, Golemi S, Maculotti P, Farina D, Maroldi R. Radiographic severity index in COVID-19 pneumonia: relationship to age and sex in 783 Italian patients. Radiol Med. 2020 May;125(5):461-464. doi: 10.1007/s11547-020-01202-1. Epub 2020 May 1. PMID 32358691